CLINICAL TRIAL: NCT00904059
Title: Open-Label, Randomized, Multiple-Dose, Drug-Drug Interaction Study to Assess the Pharmacokinetics and Safety of BMS-790052 and BMS-650032 Co-administered in Healthy Subjects
Brief Title: Drug-Drug Interaction Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AI447-009
Record Dates: First submitted 2009-04-21; First posted 2009-05-19 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Group A (Experimental)
  Interventions: Drug: BMS-650032
- Treatment Group B (Experimental)
  Interventions: Drug: BMS-790052
- Treatment Group C (Experimental): Treatment Groups A and B are followed by Treatment Group C: A combination of BMS-650032 (200 mg) and BMS-790052 (30 mg)
  Interventions: Drug: BMS-650032; Drug: BMS-790052

INTERVENTIONS:
Drug: BMS-650032 — Capsules, Oral, 600 mg, Q12h, Days 1-7
  Arms: Treatment Group A
Drug: BMS-790052 — Capsules, Oral, 60 mg, Q24h, Days 1-7
  Arms: Treatment Group B
Drug: BMS-650032 — Capsules, Oral, 200 mg, Q12h, Days 8-21
  Arms: Treatment Group C
Drug: BMS-790052 — Capsules, Oral, 30 mg, Q24h, Days 8-21
  Arms: Treatment Group C

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and safety of BMS-790052 and BMS-650032 when co-administered and when administered alone

DETAILED DESCRIPTION:
Pharmacokinetics and Safety in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 49 years
* Females who are not of childbearing potential, pregnant or breastfeeding
* Subject Body Mass Index (BMI) of 18 to 32 kg/m²

Exclusion Criteria:

* Women of child bearing potential
* Male subjects who have sex with women who are unwilling to agree to practice male barrier contraception during study participation and for a least 12 weeks following dosing
* Any significant acute or chronic medical illness
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
* Prior exposure to BMS-650032 or BMS-790052
* Positive for HIV or HCV

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters including AUC (TAU) Cmax and Cmin | Day 21 pharmacokinetic assessment

SECONDARY OUTCOMES:
To assess the safety, tolerability, and fractional excretion of sodium when BMS-709952 and BMS-650032 are co-administered | Within 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx